CLINICAL TRIAL: NCT02904005
Title: National Multicentric Study on the Predictive Factors for Suicidal Behavior During a Major Depressive Episode
Brief Title: Predictors of Suicidal Behavior in Depression
Acronym: SECS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Lille (Other); Centre Hospitalier Universiatire La Conception, Marseille (Unknown); Centre Hospitalier Régional et Universitaire de Brest (Other); Hôpital Saint Anne, Paris (Unknown); Créteil Hospital (Other); Centre Hospitalier Charles Perrens, Bordeaux (Other Government); Centre Hospitalier Universiatire Lyon (Unknown); Centre Hospitalier Universitaire de Nīmes (Other); INSERM U1061 Montpellier (Unknown); Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UF 9475; 2014-A01316-41 (Other: Agence Nationale de sécurité des Médicaments)
Record Dates: First submitted 2016-07-19; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-07

CONDITIONS: Suicidal Behavior; Depression; Traumatic Events; Impulsivity Aggression
Keywords: Suicide; Prediction; Prospective study; Suicide attempt; Risk management
MeSH Terms: conditions — Depression; Suicide; Suicide, Attempted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Depressed patients (Other): Depressed patients with a recent suicide attempt or without any personal history of suicide attempt
  Interventions: Other: Standardized assessment on depressed patients

INTERVENTIONS:
Other: Standardized assessment on depressed patients — At inclusion, socio-demographic characteristics, main life events, psychopathology (comorbidity, personality dimensions, characterisation of SB) and biological sample will be performed by psychiatrist and nurse. Investigators will retrieve the results of biological assays routinely made as part of standard collect biological results routinely done for all depressed patient.
  At follow-up (3 months, 6 months, 12 months), they will assess thymic state, occurrence of suicidal ideation and suicide attempt and environmental stressors. In case of non response, the general physician or the psychiatrist in charge of the patient will be contacted to assess the occurrence of SB during the year. In case of death or absence of clinical information, a request for cause of death certificate will be carried out through tne National Institute of Health and Medical research (INSERM) Unit 1018 / Epidemiological center on medical causes of death (CépiDc).

SUMMARY:
This study aims at identifying predictors of suicidal behaviors in depressed subjects. Investigators will first compare demographic, clinical, and biological features of depressed recent suicide attempters (within one week) and depressed subjects without lifetime history of suicide attempt. Baseline risk factors for suicide will be used to predict the risk of attempting suicide during a one year follow-up. A thorough evaluation of these patients will allow to identify the factors associated with suicidal risk and develop a simplified risk score that could be used in clinical settings to improve our practice.

DETAILED DESCRIPTION:
Background and rationale:

Suicidal behavior (SB) is a major health problem in France, with more than 10,000 suicides (6th UE28) and 220 000 suicide attempts (SA) per year. A large percentage of men (6%) and women (9%) in France have made at least one SA. Moreover, suicide is the second leading cause of death among the youngest (15-44 years). The clinical model currently admitted for understanding SB is a stress vulnerability model. But to date, scientists have not (yet) a clinical application for the research on SB. The management of psychiatric patients, including depressed subjects, faces the impossibility of detecting those at high risk of occurrence of SB. Indeed, although many risk factors for SB are known, their predictive value is very low. In addition, these risk factors are primarily derived from cross-sectional studies. The identification of predictors, using a standardized evaluation would allow clinicians to identify the subject at high risk of SB for which therapeutic interventions and the organization of care should be particularly aggressive and intensive.

Objectives:

Main objective: To identify predictors (clinical, biological, environmental) of the occurrence of SB during 12 months in a population of depressed suicide attempters and lifetime non attempters to optimize a short standardized evaluation applicable to emergency settings.

Secondary objectives: 1) To build a multidimensional score for predicting the risk of recurrence of suicide attempt among suicide attempters ; 2) To evaluate the prospective performance of this score to predict emergence of suicide attempt among depressed patients without history of suicide attempt; 3) To identify predictors of suicidal spectrum (suicidal thoughts, suicidal planification, suicide attempt and completed suicide) in depressed subjects ; 4) To evaluate the feasibility of a multicenter network that will use standardized assessments to evaluate suicidal risk through a secured website.

Methods:

2000 patients with major depressive episode will be recruited in the emergency departments and post-acute care units of 14 French hospitals, and then will be followed for 12 months. For every depressed patient admitted within 48 hours of a suicide attempt (case), a depressed patient without lifetime personal history of SB (psychiatric control) will be included. Cases will be mainly recruited in emergency settings; psychiatric controls will be mainly recruited from the inpatient units (hospital stay <7 days) and outpatient units to limit selection bias.

At inclusion, at 3, 6 and 12 months, clinical and biological assessments will ne realized.

Statistical analyses:

1) Kaplan-Meier and Cox models adjusted for potential confounding factors, 2) Univariate and multivariate analysis, 3) Establishment of a predictive score from multivariate analyses.

Short-term perspectives:

1) Optimization of standardized assessment of suicidal risk in depressed patients applicable in daily practice, and 2) Development of a network of clinical centers involved in suicidology field to promote specific care and research.

Long-term perspectives:

1) Access to a computerized assessment tool via the Internet to improve the management of depressed patients all over France 2) Understanding of the psychological and biological factors underlying SB in the context of mood disorders, and 3) Development of preventive and therapeutic approaches.

ELIGIBILITY:
Inclusion criteria:

* >18 years old
* Diagnostic Statistical Manuel IV (DSM IV) criteria for major depressive episode (
* Subject signs a non-opposition form
* Able to understand the nature, purpose and methodology of the study
* Affiliated with a French social security agency
* Not planning to change residence within 12 months
* Available by phone and / or email

Specific inclusion criteria for the suicide group:

- Admission to the hospital within 48 hours of the last suicide attempt.

Specific inclusion criteria for emotional control group:

- No history of lifetime suicide attempt suicide.

Exclusion criteria:

* Patients hospitalized for more than 7 days
* Refusal to participate
* Individual deprived of freedom (by judicial or administrative decision)
* Individual protected by law (guardianship)
* Subject to exclusion period in another protocol
* Not affiliated to a social security agency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Suicide attempt during follow-up | At one year
  Evaluation of the occurrence of a suicide attempt by the Columbia-Suicide Severity Rating Scale (C-SSRS )

SECONDARY OUTCOMES:
Depressive level | At 3, 6 and 12 months after the inclusion
  Measured by clinician with Inventory of Depressive Symptomotology (IDS-C 30)
Depressive level | At 3, 6 and 12 months after the inclusion
  Measured with a self questionnaire Quick Inventory of Depressive Symptomatology (QIDS-RS)
Anxiety | At 3, 6 and 12 months after the inclusion
  Measured with a self questionnaire the State-Trait Anxiety Inventory (STAI)

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No